CLINICAL TRIAL: NCT03333408
Title: Determining the Necessity for Postoperative Antibiotics After Salivary Stent Placement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Our Lady of the Lake Hospital (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LSUHSC-IRB 9908
Record Dates: First submitted 2017-10-20; First posted 2017-11-06 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Salivary Duct
MeSH Terms: interventions — Clindamycin; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Antibiotic) (Active Comparator): Group A will receive postoperative oral antibiotics for 10 - 14 days (Clindamycin or Augmentin) upon discharge.
  Interventions: Drug: Postoperative Oral Antibiotics (Clindamycin or Augmentin)
- Group B (no Antibiotic) (No Intervention): Group B will not be given postoperative oral antibiotics upon discharge.

INTERVENTIONS:
Drug: Postoperative Oral Antibiotics (Clindamycin or Augmentin) — Patients will receive postoperative oral antibiotics (Clindamycin or Augmentin) for 10-14 days upon discharge.
  Arms: Group A (Antibiotic)

SUMMARY:
Salivary duct stent placement is a common practice to maintain duct patency after salivary duct repair or interventional sialoendoscopy; procedures performed to manage salivary duct pathology such as stenosis, traumatic injury or most commonly salivary duct stones. It is common practice for patients to receive perioperative antibiotics while undergoing interventional sialoendoscopy and postoperative oral antibiotic therapy with Clindamycin or Augmentin for 10-14 days, if a short term (2 week) salivary duct stenting was considered necessary due to the nature of the intervention. However, In reviewing the literature, there are controversial trials that indicate post-operative antibiotics may not be best practice in all surgical scenarios, as the adverse events ie. gastrointestinal disturbances, nausea, Clostridium difficile (C.diff) infection and antibiotic resistance over time surrounding overuse of antibiotics may outweigh the clinical need for the antibiotic regiment and the chances of post-operative infection.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (18 years of age or older) who are undergoing salivary duct surgery and stent placement at Our Lady of the Lake Regional Medical Center

Exclusion Criteria:

* Patients who are unwilling to consent to the study and/or to being placed in a randomized arm of either receiving post-operative antibiotics or not receiving post-operative antibiotics
* Patients with acute infections at the time of surgery
* Patients who are immunocompromised
* Patients who are recruited but then have early dislodgement of the stent
* Patients who do not complete their postoperative antibiotic therapy due to intolerance or antibiotic side effects. However, data on these patients will be recorded to provide an observational results that will support the need for this investigation on antibiotic use.
* Patients who are in the non-post operative antibiotic arm but choose to put themselves on antibiotics without consultation from the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative infection | 2 weeks
  The primary endpoint will be the determination of clinical infection between the time points post-operation to the 2 week follow-up visit when the stent is removed as indicated by evidence of purulence or erythema at the surgical site, fever and elevated white blood cell count.

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Walvekar, M.D., Principal Investigator — Our Lady of the Lake Hospital
Locations (1):
- Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang MS, Gonzalez ML, Dodson TB. Do Antibiotics Decrease the Risk of Inflammatory Complications After Third Molar Removal in Community Practices? J Oral Maxillofac Surg. 2017 Feb;75(2):249-255. doi: 10.1016/j.joms.2016.09.044. Epub 2016 Oct 6. PMID 28341449
- [Background] Taub D, Yampolsky A, Diecidue R, Gold L. Controversies in the Management of Oral and Maxillofacial Infections. Oral Maxillofac Surg Clin North Am. 2017 Nov;29(4):465-473. doi: 10.1016/j.coms.2017.06.004. Epub 2017 Aug 18. PMID 28823889
- [Background] Fleming-Dutra KE, Hersh AL, Shapiro DJ, Bartoces M, Enns EA, File TM Jr, Finkelstein JA, Gerber JS, Hyun DY, Linder JA, Lynfield R, Margolis DJ, May LS, Merenstein D, Metlay JP, Newland JG, Piccirillo JF, Roberts RM, Sanchez GV, Suda KJ, Thomas A, Woo TM, Zetts RM, Hicks LA. Prevalence of Inappropriate Antibiotic Prescriptions Among US Ambulatory Care Visits, 2010-2011. JAMA. 2016 May 3;315(17):1864-73. doi: 10.1001/jama.2016.4151. PMID 27139059
- [Background] Dhiwakar M, Clement WA, Supriya M, McKerrow W. Antibiotics to reduce post-tonsillectomy morbidity. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD005607. doi: 10.1002/14651858.CD005607.pub4. PMID 23235625
- [Background] Aljfout Q, Alississ A, Rashdan H, Maita A, Saraireh M. Antibiotics for Post-Tonsillectomy Morbidity: Comparative Analysis of a Single Institutional Experience. J Clin Med Res. 2016 May;8(5):385-8. doi: 10.14740/jocmr2523w. Epub 2016 Mar 20. PMID 27081424
- [Background] Santana RS, Viana Ade C, Santiago Jda S, Menezes MS, Lobo IM, Marcellini PS. The cost of excessive postoperative use of antimicrobials: the context of a public hospital. Rev Col Bras Cir. 2014 May-Jun;41(3):149-54. doi: 10.1590/s0100-69912014000300003. English, Portuguese. PMID 25140644
- [Background] Chen S, Le CH, Liang J. Practice patterns in endoscopic dacryocystorhinostomy: survey of the American Rhinologic Society. Int Forum Allergy Rhinol. 2016 Sep;6(9):990-7. doi: 10.1002/alr.21759. Epub 2016 Apr 6. PMID 27060784
- [Background] Araujo da Silva AR, Albernaz de Almeida Dias DC, Marques AF, Biscaia di Biase C, Murni IK, Dramowski A, Sharland M, Huebner J, Zingg W. Role of antimicrobial stewardship programmes in children: a systematic review. J Hosp Infect. 2018 Jun;99(2):117-123. doi: 10.1016/j.jhin.2017.08.003. Epub 2017 Aug 12. PMID 28807835
- [Background] Stultz JS, Doern CD, Godbout E. Antibiotic Resistance in Pediatric Urinary Tract Infections. Curr Infect Dis Rep. 2016 Dec;18(12):40. doi: 10.1007/s11908-016-0555-4. PMID 27761778
- [Background] Phuong NTK, Hoang TT, Van PH, Tu L, Graham SM, Marais BJ. Encouraging rational antibiotic use in childhood pneumonia: a focus on Vietnam and the Western Pacific Region. Pneumonia (Nathan). 2017 Apr 25;9:7. doi: 10.1186/s41479-017-0031-4. eCollection 2017. PMID 28702309
- [Background] Linder JA. Editorial commentary: antibiotics for treatment of acute respiratory tract infections: decreasing benefit, increasing risk, and the irrelevance of antimicrobial resistance. Clin Infect Dis. 2008 Sep 15;47(6):744-6. doi: 10.1086/591149. No abstract available. PMID 18694343